CLINICAL TRIAL: NCT02850770
Title: Phone Messaging for Physical Activity and Social Support Prompting Among Low-Income Latino Patients: A Randomized Pilot Study
Brief Title: Physical Activity and Social Support Prompting Via Phone Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Los Angeles County Department of Public Health (Other Government)
Responsible Party: Principal Investigator, Shinyi Wu, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS-13-00471; 3U54NS081764-03S1 (NIH)
Record Dates: First submitted 2016-04-12; First posted 2016-08-01 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Other): Pedometers and walking logs
  Interventions: Behavioral: Pedometers and Walking Logs
- Phone Messaging (Experimental): Phone Messaging
  Interventions: Behavioral: Pedometers and Walking Logs; Behavioral: Phone Messaging
- Phone Messaging + Family/Friend Support (Experimental): Phone Messaging + Family/Friend Support
  Interventions: Behavioral: Pedometers and Walking Logs; Behavioral: Phone Messaging; Behavioral: Family/Friend Support

INTERVENTIONS:
Behavioral: Pedometers and Walking Logs — Participants were recommended to use the pedometer and walking log to self-monitor how many steps participants walked each day. Participants were recommended to gradually increase daily steps over the course of 12 weeks until reaching 10,000 steps per day. Participants were also recommended to walk at a brisk pace for 3000 of these steps, which roughly translates to 30 minutes per day.
Behavioral: Phone Messaging — Participants received short text or voice messages (depending on participant preference) as reminders to review daily step goals and to self-monitor; explaining the benefits of regular physical activity, importance of regular physical activity to daily life, and ways to overcome commonly identified barriers to physical activity; asking participants to report on their physical activity performance; providing feedback based on responses.
  Arms: Phone Messaging; Phone Messaging + Family/Friend Support
Behavioral: Family/Friend Support — Participants identified a family member or close friend (FF) to receive short text or voice messages (depending on FF preference) with suggested behaviors that are perceived as supportive by individuals making physical activity behavior changes.
  Arms: Phone Messaging + Family/Friend Support

SUMMARY:
The objective of this study was to investigate the feasibility, perceived usefulness, and potential effectiveness of a short text or voice message intervention to activate 1) physical activity behavior change among low-income, urban, Latino patients in diabetes management and 2) supportive behaviors by family members or close friends.

DETAILED DESCRIPTION:
Despite the promise of phone-based interventions to effectively support diabetes self-management (DSM), little is known about their impact on the outcomes of highly vulnerable populations such as low-income, inner-city, racial/ethnic minorities. And while phone-based interventions have generally been successful at reaching and engaging adults with diabetes, they have failed to do the same with family members/friends (FF) whom are a promising source of ongoing support for DSM. The objective of this study was to investigate the feasibility, perceived usefulness, and potential effectiveness of a short text or voice message (ST/VM) intervention to activate 1) physical activity (PA) behavior change among low-income, urban, Latino patients in diabetes management and 2) supportive behaviors by FF. The investigators conducted a 12-week pilot study in which participants were randomized into one of three study arms: control, phone messaging (PM), and phone messaging plus social support from FF (PM+FF). Participants were recruited in person from a diabetes management program at a safety-net ambulatory care clinic. All participants were given a pedometer and walking log for self-monitoring. Participants in the PM and PM+FF arms received ST/VMs as reminders to review daily step goals and to self-monitor; explaining the benefits of regular PA, importance of regular PA to daily life, and ways to overcome commonly identified barriers to PA; asking participants to report on PA performance; providing feedback based on responses. Participants in the PM+FF identified a FF to receive ST/VMs with suggested behaviors that are perceived as supportive by individuals making PA behavior changes. Participants received semi-structured assessments in person at baseline, 6 weeks, and 12 weeks. Participants were asked about the extent to which the program enhanced the participant's ability to make PA behavior changes. The primary outcome measures were daily step counts and perceived FF social support.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Diagnosis of type 2 diabetes
* No medical conditions restricting patient from beginning a walking program
* Preferred language of English or Spanish, self-identifies as a Hispanic
* Ability to walk without the use of assistive devices such as canes or walkers
* Available to attend three interviews at the clinic
* Does not plan to move away from the region or be out of the country during the next three months
* Has a working phone where they can receive regular short text or voice messages for three months

Exclusion Criteria:

* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in average daily steps assessed by pedometers | Baseline, 6 weeks, 12 weeks
  Change in average daily steps assessed using pedometer 7-day data storage

SECONDARY OUTCOMES:
Change in body mass index | Baseline, 6 weeks, 12 weeks
  Change in Body Mass Index, which was calculated as weight (in kilograms) over height squared (in centimeters)
Change in exercise self-efficacy assessed using the Exercise Self-Efficacy Scale | Baseline, 6 weeks, 12 weeks
  Change in exercise self-efficacy assessed using the Exercise Self-Efficacy Scale
Change in barriers self-efficacy assessed using the Barriers Self-Efficacy Scale | Baseline, 6 weeks, 12 weeks
  Change in barriers self-efficacy assessed using the Barriers Self-Efficacy Scale
Change in perceived family/friend social support assessed using the Social Support and Exercise Survey | Baseline, 6 weeks, 12 weeks
  Change in perceived family/friend social support assessed using the Social Support and Exercise Survey

OTHER OUTCOMES:
Change in perceived usefulness assessed using patient interviews | 6 weeks, 12 weeks
  At the 6- and 12-week follow-up interviews, participants were asked a series of unstructured questions regarding the extent to which the program enhanced a participant's ability to make physical activity behavior changes. These questions inquired about participants' thoughts on setting PA goals, self-monitoring, educational and feedback ST/VMs, and the idea of using ST/VMs to communicate with patients about PA behavior change. For participants in the PM+FF arms, the questions also inquired about supportive behaviors exhibited by FF since the start of the program and participants' thoughts on the idea of using ST/VMs to communicate with FF about patients' PA behavior changes. Investigators also asked if participants would be willing to participate in a similar program in the future and if participants would be willing to recommend the program to other patients. The latter two were yes/no questions.
Change in perceived usability of pedometers assessed via patient interviews | Baseline, 6 weeks, 12 weeks
  Semi-structured patient interview questions inquiring about the degree to which participants perceived the pedometers to be easy to use
Change in perceived barriers to receipt of and engagement with ST/VMs assessed via patient interviews | 6 weeks, 12 weeks
  Semi-structured patient interview questions inquiring about participants' perceived barriers to the receipt of and engagement with ST/VMs
Change in engagement with ST/VMs requiring a response assessed via call logs | 6 weeks, 12 weeks
  Percentage of times that participants responded to ST/VMs requiring a response
Change in receipt of ST/VMs assessed via self-report and call logs | 6 weeks, 12 weeks
  Percentage of short text messages delivered that were received assessed via self-report, and percentage of voice messages that were received assessed via call logs
Change in non-compliance with wearing pedometer assessed via pedometer and walking log | Baseline, 6 weeks, 12 weeks
  Percentage of patients that did not wear the pedometer for a minimum of three consecutive days for at least 10 hours per day. This data will be obtained using the pedometer 7-day memory storage and participants' self-reported hours of use.
Recruitment and retention rates assessed via recruitment and follow-up logs | 1 day (Recruitment), 6 weeks, 12 weeks
  Percentage of patients that were screened, were eligible to participate, and enrolled in the study. Percentage of patients who completed the 6-week and 12-week follow-up assessments.
Sufficiency or restrictiveness of eligibility criteria assessed via recruitment logs | 1 day (Recruitment)
  Percentage of patients that were screened, but were ineligible to participate and the reasons why

CONTACTS AND LOCATIONS:
Overall Officials: Shinyi Wu, Ph.D., Principal Investigator — University of Southern California

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ramirez M, Wu S. Phone Messaging to Prompt Physical Activity and Social Support Among Low-Income Latino Patients With Type 2 Diabetes: A Randomized Pilot Study. JMIR Diabetes. 2017 Jun 6;2(1):e8. doi: 10.2196/diabetes.7063. PMID 30291094